CLINICAL TRIAL: NCT01888276
Title: Study of Words Generation in Compulsives Gamblers and Healthy Volunteers: Comparison With a Study of Parkinson's Disease Patients
Brief Title: Words Generation in Compulsives Gamblers and Parkinson's Disease Patients
Acronym: FLUENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11 225 02
Record Dates: First submitted 2012-02-20; First posted 2013-06-27 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson Disease
Keywords: Words generation, compulsive gamblers
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy volunteers (Other): evaluation of word generation and of motivation
  Interventions: Other: evaluation of word generation and of motivation
- compulsive gamblers (Other): evaluation of word generation and of motivation
  Interventions: Other: evaluation of word generation and of motivation

INTERVENTIONS:
Other: evaluation of word generation and of motivation — Each subject will realize twice each test during 2 sessions with one hour in between :
  During the session 1 :
  * The test of words generation, which is to produce action verbs in response to 40 nouns, and noun in response to verbs.
  * The test of Stroop that assesses selective attention
  During the session 2:
  * The test of words generation, which is to produce action verbs in response to 40 nouns, and noun in response to verbs.
  * The task of the casino (Iowa Gambling Test)
  * The task of landing
  * The test of Stroop

SUMMARY:
The pathophysiology of compulsive disorders as gambling could be close to behavior problems encountered in Parkinson's disease associated with a hyperactivity of the motivational system.

Thanks to the words generation test, which reflects the cortico-subcortical loop functioning, involved in motivation, we want to evaluate and compare using tools (words generation and behavioral tests) the motivational functioning of gamblers and healthy volunteers that we can then compare to that of Parkinson's patients with and without behavioral hyperdopaminergic disorders which were explored in another study.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate performance during words generation in gamblers and healthy volunteers compare to those of PD patients with and without hyper-dopaminergic behaviors collected during another study.

2 groups of subjects will be recruited for the study: 20 compulsive gamblers and 20 healthy volunteers

Each subject will realize twice each test during 2 sessions with one hour in between :

During the session 1 :

* The test of words generation, which is to produce action verbs in response to 40 nouns, and noun in response to verbs.
* The test of Stroop that assesses selective attention

During the session 2:

* The test of words generation, which is to produce action verbs in response to 40 nouns, and noun in response to verbs.
* The task of the casino (Iowa Gambling Test)
* The task of landing
* The test of Stroop

We supposed that the performance of compulsive gamblers in words generation test will be higher than those of healthy volunteers, themselves superior to those of PD patients with a hyper-dopaminergic behavior, themselves superior to those of PD patient without hyper-dopaminergic behavior.

ELIGIBILITY:
Inclusion Criteria:

For healthy volunteers :

* Subject from 30 to 75 years old (Male and female)
* Subject with French mother tongue
* Subject who give their informed and signed consent.
* Subject affiliated to a social protection program

For compulsive gamblers :

* Subject from 30 to 75 years old (Male and female)
* Subject with French mother tongue
* Subject with at least 5 criteria of 10 DSM IV diagnostic criteria for pathological gambling
* Subject who give their informed and signed consent.
* Subject affiliated to a social protection program

Exclusion Criteria:

For healthy volunteers and compulsive gamblers :

* Presence of apathy defined as a score greater or equal to 14 on the scale of Starkstein
* Presence of severe depression defined as a score greater or equal to 25 on the scale BDI (Beck Depression Inventory)
* Presence of dementia defined as a score below 25 on the MMSE
* Subject with vision problems making it impossible for the tests
* Pregnant women
* Subject under tutelage, curatelle or law protection
* Subject included in an other clinical study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Changement of number of mistake during the words generation test | one hour

SECONDARY OUTCOMES:
changement of number of uncorrected errors during the Stroop test which reflects the incapacity to inhibit the reading and that evaluates attention | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Christine Brefel, MD, Principal Investigator — UH Toulouse
Locations (1):
- CHU toulouse, Toulouse, France